CLINICAL TRIAL: NCT00859651
Title: Effects of High-Dose Vitamin D on Circulating Vitamin D Levels and Breast Density in Postmenopausal Women at High Risk for Breast Cancer Development
Brief Title: Vitamin D in Postmenopausal Women at High Risk for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Avon Foundation (Other)
Responsible Party: Principal Investigator, Katherine D. Crew, Associate Professor of Medicine and Associate Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAD3638
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Results first posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: breast cancer chemoprevention; vitamin D; breast density
MeSH Terms: conditions — Breast Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 20,000 IU weekly (Active Comparator): Postmenopausal women who are at increased risk for breast cancer development receiving vitamin D3, oral cholecalciferol 20,000 IU weekly, for one year.
  Cholecalciferol 20,000 IU (2 active capsules + 1 matching placebo capsule)
  Interventions: Drug: Cholecalciferol; Drug: Placebo capsule
- 30,000 IU weekly (Active Comparator): Postmenopausal women who are at increased risk for breast cancer development receiving vitamin D3, oral cholecalciferol 30,000 IU weekly, for one year.
  Cholecalciferol 30,000 IU (3 active capsules)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Cholecalciferol is a vitamin D3. Vitamin D is important for the absorption of calcium from the stomach and for the functioning of calcium in the body. Cholecalciferol is used to treat or prevent many conditions caused by a lack of vitamin D.
  Cholecalciferol will be available in gel capsule form at 10,000 IU (0.25 mg cholecalciferol) each.
  Other Names: Vitamin D3
Drug: Placebo capsule — Matching placebo capsules
  Other Names: Placebo
  Arms: 20,000 IU weekly

SUMMARY:
This is a phase II study which will enroll 20 postmenopausal women who are at high risk for breast cancer development. The goal is to determine whether a one-year intervention of high-dose vitamin D at 2 different doses (20,000 IU weekly or 30,000 IU weekly) will increase circulating blood levels of vitamin D and to obtain preliminary data on the biologic effects of vitamin D for breast cancer prevention.

DETAILED DESCRIPTION:
Participants will receive oral vitamin D3, cholecalciferol 20,000 IU or 30,000 IU weekly. Before beginning the intervention, the participants will have a general physical exam including a clinical breast exam and anthropometric measures, a morning blood draw (for analysis of 25(OH)D, 1,25(OH)D, parathyroid hormone (PTH), insulin-like growth factor (IGF)-I, insulin-like growth factor-binding protein 3 (IGFBP-3), estradiol, estrone, testosterone, and sex hormone-binding globulin (SHBG) at baseline, 6 months, and 12 months) and a bilateral mammogram (at baseline and 12 months). Participants will also complete a baseline questionnaire, collecting data on demographic information and breast cancer risk factors. In addition, we will be collecting data on vitamin D sources from diet and sunlight exposure using a validated questionnaire administered at baseline and 12 months.

For follow-up visits, the participant will be seen at the study site at months 3, 6, 9, and 12. During these visits, drug will be dispensed, adherence ascertained, and adverse events will also be assessed. In addition, blood (serum calcium, albumin, creatinine) and urine (urine calcium, creatinine) will be collected to monitor for toxicity. A 24-hour urine collection will be conducted at baseline and 12 months to assess for hypercalciuria. After the 1 year intervention, all participants will have a complete physical exam including clinical breast exam, a bilateral mammogram, blood draw, and complete a follow-up questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Elevated risk of breast cancer defined as having at least one of the following: (1) Predicted 5-year modified Gail model risk of 1.67% or greater, (2) Lobular carcinoma in situ, (3) Known BRCA1 or BRCA2 deleterious mutation carrier, (4) Prior history of ductal carcinoma in situ, if no current tamoxifen use or prior radiation to the contralateral breast.
* Age 21 years or older.
* Postmenopausal defined as > 6 months since the last menstrual period, prior bilateral oophorectomy, or serum follicle-stimulating hormone (FSH)/luteinizing hormone (LH) values consistent with institutional normal values for the postmenopausal state.
* Baseline mammographic density ≥25% as assessed qualitatively by the mammographer (25-50% = "scattered fibroglandular densities"; >50-75% = "heterogeneously dense breasts"; >75% = "extremely dense breasts").
* Baseline serum 25-hydroxyvitamin D <32 ng/ml.
* Normal breast exam and mammogram (Breast Imaging Reporting and Data System (BIRADS) score of 1 or 2) or abnormal breast imaging with a benign breast biopsy without evidence of cancer. Normal baseline breast magnetic resonance imaging (MRI) (BIRADS score of 1, 2, or 3).
* Prior tamoxifen or raloxifene use is allowed provided treatment is discontinued at least 28 days prior to enrollment.
* At least one breast available for imaging. No bilateral breast implants.
* Willingness to not take vitamin D supplements during the one year intervention, but up to 1000mg of calcium supplementation is allowed.
* Normal serum calcium.
* Adequate renal and hepatic function: serum creatinine, bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase < 2.0 x the institutional upper limit of normal (IULN).
* Performance status of 0 or 1.

Exclusion Criteria:

* Other prior malignancy. The following is allowed: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the participant is currently in complete remission, or any other cancer (including breast cancer) for which the participant has been disease-free for 5 years.
* History of kidney stones.
* Hypersensitivity reactions to vitamin D.
* On estrogen replacement therapy.
* Significant medical or psychiatric condition that would preclude study completion.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine D Crew, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data for this study (NCT00859651; n=20 postmenopausal; 8 received 20,000 IU/week and 12 received 30,000 IU/week) is combined with the data for another study (NCT00976339; n=20 premenopausal; 10 received 20,000 IU/week and 10 received 30,000 IU/week). Resulting in a combination of 18 receiving 20,000 IU/week and 22 receiving 30,000 IU/week.
Groups:
- Cholecalciferol 20,000 IU Group: Postmenopausal women who are at increased risk for breast cancer development receiving vitamin D3, oral cholecalciferol 20,000 IU weekly, for one year.
- Cholecalciferol 30,000 IU Group: Postmenopausal women who are at increased risk for breast cancer development receiving vitamin D3, oral cholecalciferol 30,000 IU weekly, for one year.
Period: Overall Study
Arm/Group | Cholecalciferol 20,000 IU Group | Cholecalciferol 30,000 IU Group
Started | 18 | 22
Completed | 18 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data for this study (NCT00859651; n=20) is combined with the data for another study (NCT00976339; n=20).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cholecalciferol 20,000 IU Group | Cholecalciferol 30,000 IU Group | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Median (Full Range); unit: years] | 50.0 [45 to 73] | 50.5 [37 to 69] | 50 [37 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum 25(OH)D
Description: 25(OH)D level at the end of one year intervention
Time Frame: Baseline to 1 year
Population: Data for this study (NCT00859651; n=20) is combined with the data for another study (NCT00976339; n=20).
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cholecalciferol 20,000 IU Group | Cholecalciferol 30,000 IU Group
Number analyzed (Participants) | 18 | 22
ng/ml | 25 (5) | 33 (9)

2. Secondary Outcome: Change in Percent Density
Description: Assessed by mammography and breast MRI.
Time Frame: Baseline to 1 year
Population: Data for this study (NCT00859651; n=20) is combined with the data for another study (NCT00976339; n=20).
Measure: Mean (Standard Deviation); unit: percentage of breast density
Arm/Group | Cholecalciferol 20,000 IU Group | Cholecalciferol 30,000 IU Group
Number analyzed (Participants) | 18 | 22
percentage of breast density | 3 (1) | 1 (1)

ADVERSE EVENTS:
Description: For the Outcome Measure data analysis, the investigator combined the data for this study (NCT00859651; n=20) with the data for another study (NCT00976339; n=20), since both studies are under the same investigational new drug (IND). Therefore, the total number of participants analyzed is 40.
Groups:
- Cholecalciferol 20,000 IU: Postmenopausal women who are at increased risk for breast cancer development receiving vitamin D3, oral cholecalciferol 20,000 IU weekly, for one year.
- Cholecalciferol 30,000 IU: Postmenopausal women who are at increased risk for breast cancer development receiving vitamin D3, oral cholecalciferol 30,000 IU weekly, for one year.
Arm/Group | Cholecalciferol 20,000 IU | Cholecalciferol 30,000 IU
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 14/18 | 22/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cholecalciferol 20,000 IU (N=18) | Cholecalciferol 30,000 IU (N=22)
Hypertension (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 1 | 6
Weight gain (Investigations) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 7
Headache (Nervous system disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 6
Diarrhea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 4
Hypercalciuria (Metabolism and nutrition disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The investigator combined the data for this study (NCT00859651; n=20) with the data for another study (NCT00976339; n=20). Therefore, the total number of participants analyzed is 40 for Outcome Measures and Adverse Events sections.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes